CLINICAL TRIAL: NCT00684749
Title: Pilot Study to Investigate The BodyLogic TM System (Mentor) in Breast Augmentation.
Brief Title: A Pilot Study to Evaluate the BodyLogic TM System (Mentor) in Augmentation Mammaplasty
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: Mentor Worldwide, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 0801E25711
Record Dates: First submitted 2008-05-22; First posted 2008-05-28 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Breast Augmentation; Breast Reconstruction
Keywords: Mentor BodyLogic TM System; Breast augmentation; Breast implant choice; Reoperation rates

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
At a national level of 15%, the reoperation rate following augmentation mammaplasty is too high. We are conducting a survey to examine the pre-operative methods by which plastic surgeons determine implant volume, size, shape and location; and to determine if the Mentor "BodyLogic"TM System can successfully improve outcomes. We will evaluate how measurements taken using "BodyLogic"TM influence choice of implant and whether there are any re-operations, particularly for size change. We hypothesize that using this system will help surgeons choose appropriate implants that will decrease the rate of reoperations, especially for size change.

DETAILED DESCRIPTION:
We are planning to survey 10 high volume plastic surgeons that perform at least 10 breast augmentations a month and to collect data on at least 300 patients. The enrollment period will be 3 months.

As part of this study, we are having the following steps performed:

1. Complete a 'general preference questionnaire', designed to document current preoperative planning and assessment methods for breast augmentation.
2. For each study patient, a pre-operative "BodyLogic"TM worksheet will be completed. Then, using the provided Implant Selection Booklet, the actual implant will be selected. The surgeon will maintain a key of the patients, and will identify them to the investigators only by subject number, and return these forms in provided stamped, self-addressed envelopes.
3. The patient returns at 1-3 months and 8-12 months for completion of the respective "Body-Logic" post-operative worksheets for each visit and the surgeon will send us the data in the provided envelopes periodically.
4. If during the course of the data collection, the surgeon has to re-operate on any patient, he/she will fill the "re-operative form" and send it to us.
5. Finally, the surgeon will complete a post-study evaluation questionnaire to help us understand how the "BodyLogic"TM System worked for him/her and how it could be improved.

ELIGIBILITY:
Inclusion Criteria:

* Female (age > 22 years)
* Cosmetic Breast Augmentation only
* Primary breast augmentation

Exclusion Criteria:

* Breast reconstruction
* Secondary breast augmentation
* <22 years of age

Min Age: 22 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients having cosmetic breast augmentation.
Sampling Method: Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2008-05; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Umar H Choudry, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Surgeons recruited their own patients in their own offices
Pre-assignment Details: as above.
Groups:
- Total Population: All surgical patients
Period: Overall Study
Arm/Group | Total Population
Started | 142
Completed | 142
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Total Population
Number analyzed (Participants) | 142
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 142
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Reoperation Rates
Description: Surgeon completed survey
Time Frame: 2 years
Population: All patients who were treated in the time period
Measure: Number; unit: participants
Arm/Group | Total Population
Number analyzed (Participants) | 142
participants | 6

2. Secondary Outcome: Patient Satisfaction With Outcome
Description: Patient completed a survey regarding outcome
Time Frame: 1 Year
Reporting Status: Not Posted

3. Secondary Outcome: Surgeon Satisfaction With Outcome
Description: Patient completedsurvey regarding outcome
Time Frame: 1 Year
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Total Population
Serious Adverse Events (participants affected / at risk) | 0/142
Other Adverse Events (participants affected / at risk) | 0/142

LIMITATIONS AND CAVEATS:
snap shot view, responder bias

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No